CLINICAL TRIAL: NCT04025242
Title: Objective Assessment of Adherence to Inhalers by COPD Patients
Status: Completed | Type: Observational
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor, Beaumont Hospital
Other Study IDs: INCA-COPD
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Objective adherence to inhaled therapy by patients with chronic obstructive pulmonary disease (COPD) has not been reported.

Objectives: To objectively quantify adherence to preventer Diskus inhaler therapy by patients with COPD with an electronic audio recording device (INCA).

Methods: This was a prospective observational study. On discharge from hospital patients were given a salmeterol/fluticasone inhaler with an INCA device attached. Analysis of this audio quantified the frequency and proficiency of inhaler use.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised with an exacerbation of COPD
* FEV1/FVC <70% or FEV1 <80%
* Age>40 years
* smoking history
* Previously prescribed fluticasone/salmeterol inhaler

Exclusion Criteria:

* No exacerbations in previous year
* Outpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to an acute hospital with exacerbation of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Actual rate of inhaler adherence | Three months post hospitalisation
  Inhaler adherence rate assessed using a mobile electronic device